CLINICAL TRIAL: NCT03048487
Title: Protein Consumption in Critically Ill Patients: A Retrospective Study
Brief Title: Protein Consumption in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 16.11.CLI
Record Dates: First submitted 2016-10-04; First posted 2017-02-09 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Critical Illness; Dietary Modification
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective study of protein intake and needs as well as outcomes in critically ill adult patients. Data will be collected for up to 7 days of ICU stay.

DETAILED DESCRIPTION:
This retrospective study of critically ill adults receiving enteral nutrition will assess the ability to meet estimated protein and energy needs via enteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years)
* Admitted to the ICU
* Administered at least one dose of enteral formula

Exclusion Criteria:

* Receiving exclusive oral or exclusive parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all patients with an ICU admission receiving enteral nutrition in a 36-month period.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Daily protein intake (from Parenteral Nutrition, Enteral Nutrition, oral diet, and medication) | Daily up to 7 days of ICU stay

SECONDARY OUTCOMES:
Enteral formula utilized (Standard, High protein, Very high protein) | Daily up to 7 days of ICU stay
Daily caloric intake (from Parenteral Nutrition, Enteral Nutrition, oral diet, and medication) | Daily up to 7 days of ICU stay
Estimated caloric needs (Kcal/day) | Daily up to 7 days of ICU stay
Method for estimating caloric needs (descriptive name of scale) calorie needs met. | Daily up to 7 days of ICU stay
Percentage of daily caloric needs met (%) calorie needs met. | Daily up to 7 days of ICU stay
Estimated protein needs (grams protein/day) | Daily up to 7 days of ICU stay
Method for estimating protein needs (descriptive name of scale) | Daily up to 7 days of ICU stay
Percentage of daily protein needs met (%) | Daily up to 7 days of ICU stay
Laboratory values (Blood Urea Nitrogen) | Daily up to 7 days of ICU stay
Laboratory values (Creatinine) | Daily up to 7 days of ICU stay
Laboratory values (Aspartate aminotransferase) | Daily up to 7 days of ICU stay
Laboratory values (Alanine transaminase) | Daily up to 7 days of ICU stay
Laboratory values (Glucose) | Daily up to 7 days of ICU stay
Laboratory values (Ammonia) | Daily up to 7 days of ICU stay
Gastrointestinal side effects observed in enterally fed patients in the ICU | Daily up to 7 days of ICU stay
Insulin use | Daily dose up to 7 days of ICU stay
Health Outcomes (Renal failure, Seizures, Encephalopathy, Hyperglycemia, Hypoglycemia) | Daily up to 7 days of ICU stay
Utilization of renal replacement therapy (Yes/No) | Daily up to 7 days of ICU stay
Utilization of medications to manage hepatic encephalopathy (lactulose) (Yes/No) | Daily up to 7 days of ICU stay
Neurocognitive status (Glasgow Coma Scale) | Daily up to 7 days of ICU stay
Presence of delirium (Yes/No) | Daily up to 7 days of ICU stay
ICU Length of Stay | Up to 90 Days
Hospital Length of Stay | Up to 90 Days
Ventilator days | Up to 90 Days
Antibiotic therapy days | Up to 90 Days
30 day readmission | Incidence up to 30 days post discharge
Death during hospitalization (Yes/No) | Through study completion, assessed an estimated 36 months
Destination for discharge (home, another acute care hospital, Long Term Acute Care, rehabilitation center, nursing home) | Through study completion, assessed an estimated 36 months
  Destination of Discharge will be assessed via chart review.
Discharge against medical advice (Yes/No) | Through study completion, assessed an estimated 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Layon, MD, FACP, Principal Investigator — Geisinger Clinic
Locations (3):
- United States (3):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Community Medical Center, Scranton, PA, Scranton, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania

IPD SHARING:
Plan to Share IPD: No